CLINICAL TRIAL: NCT01025154
Title: Clofarabine, Idarubicin, and Cytarabine Combination as Induction Therapy for Younger Patients With Acute Myeloid Leukemia (AML)
Brief Title: Clofarabine, Idarubicin, and Cytarabine Combination in Acute Myeloid Leukemia (AML) Induction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0431
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; AML; chemotherapy-naïve; Clofarabine; Clofarex; Clolar; Idarubicin; Idamycin; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Clofarabine; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine, Cytarabine + Idarubicin (Experimental): Induction Cycle: Clofarabine 20 mg/m^2 intravenous (IV) daily for 5 days; Idarubicin 10 mg/m^2 IV daily for 3 days; Cytarabine 1 g/m^2 IV daily for 5 days
  Interventions: Drug: Clofarabine; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Clofarabine — Induction Cycle: 20 mg/m^2 IV over approximately 1 hour daily for 5 days (days 1-5)
  Other Names: Clofarex; Clolar
Drug: Idarubicin — Induction Cycle: 10 mg/m^2 IV over approximately 30 minutes daily for 3 days (days 1-3), following clofarabine by 1 to 2 hours
  Other Names: Idamycin
Drug: Cytarabine — Induction Cycle: 1 g/m^2 IV over approximately 2 hours daily for 5 days (days 1-5), follow clofarabine by 3 to 6 hours.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride

SUMMARY:
The goal of this clinical research study is to learn if the combination of clofarabine, cytarabine, and idarubicin can help to control Acute Myeloid Leukemia (AML) in patients who are between the ages of 18 and 60 years old. The safety of this study drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Clofarabine is designed to interfere with the growth and development of cancer cells.

Idarubicin is designed to cause breaks in DNA (the genetic material of cells) of cancer cells and interfere with their growth and development.

Cytarabine is designed to insert itself into DNA of cancer cells and stop the DNA from repairing itself.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drug combination over 1 or 2 "Induction Cycles" of treatment. Whether or not you receive a second Induction Cycle depends on the disease's response to the first Induction Cycle. Each Induction Cycle will last about 4-6 weeks, depending on your reaction to the study drugs. During each Induction Cycle, you will receive the study drugs by the following schedule:

* Clofarabine, by vein, over 1-2 hours on Days 1-5.
* Cytarabine, by vein, over 2-3 hours on Days 1-5.
* Idarubicin, by vein, over about 30-60 minutes on Days 1-3.

If the disease shows a response to the treatment during the Induction Cycle(s), you may continue to receive up to 6 "Consolidation Cycles" of treatment. Each Consolidation Cycle will last about 3-10 weeks, depending on your reaction to the study drugs. During each Consolidation Cycle, you will receive the study drugs by the following schedule:

* Clofarabine, by vein, over 1-2 hours on Days 1-3.
* Cytarabine, by vein, over 2-3 hours on Days 1-3.
* Idarubicin, by vein, over 30-60 minutes on Days 1-2.

Study Visits:

On Day 1 of every cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.

Throughout the study, you will have blood and bone marrow tests to check the status of the disease and to help the doctor decide if you need additional cycles of treatment. Blood (about 1-2 tablespoons each time) will be drawn 2 times each week for routine tests during the Induction Cycles. This blood will also be drawn every week during the Consolidation Cycles.

About 3 weeks after you first receive the study drugs, you will have a bone marrow aspirate to check the status of the disease. After that, you will have a bone marrow aspirate every 2 weeks (or more often if your doctor thinks it is needed). However, if the routine blood tests show that there is still leukemia present, these bone marrow samples may not need to be collected.

You will need to stay in Houston for up to the first 5 weeks of treatment. After that, you will need to return to Houston to receive treatment, but you can have check-up visits and blood tests with your local doctor in between treatments.

Length of Study:

You will be able to receive the study drugs for up to 8 cycles (a maximum of 2 induction cycles and 6 consolidation cycles). You will be taken off study if the disease gets worse or you experience any intolerable side effects.

Follow-up Scan:

Within 8 weeks after you have stopped taking the study drug, you will have an echocardiogram or a Multiple gate acquisition scan (MUGA) scan to check your heart function.

This is an investigational study. Cytarabine and idarubicin are both FDA approved and commercially available for the treatment of patients with AML. Clofarabine is FDA approved and commercially available for the treatment of patients with acute lymphoblastic leukemia (ALL). The use of this drug combination for the treatment of AML is investigational.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML (World Health Organization (WHO) classification)
2. Patients must be chemotherapy-naïve, i.e. not have received any prior cytotoxic chemotherapy for AML (with the exception of hydroxyurea). They could have received prior therapy with hypomethylating agents, targeted, or biological agents.
3. Age 18 to 60 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
5. Serum creatinine </= 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73m^2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73m^2)=186 * (serum creatinine)^-1.154 x (age in years)^-0.023 * (0.742 if patient is female) * (1.212 if patient is black), where SCr is serum creatinine measured in mg/dL. serum bilirubin </= 1.5 * upper limit of normal (ULN) (unless increase is due to hemolysis or a congenital disorder); serum transaminases (SGPT and/or SGOT) </= 2.5 * ULN.
6. Cardiac ejection fraction >/= 45% (by either echocardiography or MUGA scan).
7. Ability to understand and provide signed informed consent.

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia (APL).
2. Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results.
3. Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, intrauterine device (IUD), diaphragm, abstinence, or condoms by their partner) over the entire course of therapy.
4. Active and uncontrolled infection requiring therapy with IV antibiotics or antifungal therapy. Prior or concurrent history of one or more opportunistic infections (e.g., cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Morita K, Kantarjian HM, Wang F, Yan Y, Bueso-Ramos C, Sasaki K, Issa GC, Wang S, Jorgensen J, Song X, Zhang J, Tippen S, Thornton R, Coyle M, Little L, Gumbs C, Pemmaraju N, Daver N, DiNardo CD, Konopleva M, Andreeff M, Ravandi F, Cortes JE, Kadia T, Jabbour E, Garcia-Manero G, Patel KP, Futreal PA, Takahashi K. Clearance of Somatic Mutations at Remission and the Risk of Relapse in Acute Myeloid Leukemia. J Clin Oncol. 2018 Jun 20;36(18):1788-1797. doi: 10.1200/JCO.2017.77.6757. Epub 2018 Apr 27. PMID 29702001
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 1/28/2010 - 2/20/2013; All participants were registered at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 63 participants registered, four (4) were excluded prior to study starting.
Period: Overall Study
Arm/Group | Clofarabine, Cytarabine + Idarubicin
Started | 59
Completed | 57
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine, Cytarabine + Idarubicin
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Overall Response: Number of Participants With Complete Remission or Complete Remission Without Platelet Recovery
Description: Overall Response (CR+CRp) defined as Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x 10^9/L and platelet count > 100 x 10^9/L, and normal bone marrow differential (< 5% blasts); and, Complete Remission without Platelet Recovery (CRp): Peripheral blood and bone marrow results as for CR, but with platelet counts of < 100 x 10^9/L. Response evaluated within 8 weeks after induction therapy.
Time Frame: 8 weeks after Induction therapy (induction cycle 4-6 weeks)
Population: Two of the fifty-nine participants were not evaluable.
Measure: Number; unit: participants
Arm/Group | Clofarabine, Cytarabine + Idarubicin
Number analyzed (Participants) | 57
participants
  Complete Remission | 42
  Complete Remission without Platelet Recovery | 3

2. Primary Outcome: Median Event-Free Survival (EFS)
Description: Event-free survival (EFS) defined as time from start of treatment to first documentation of disease relapse or death. Bayesian time-to-event model will be used to monitor progression free survival.
Time Frame: 2 years
Population: Two of the fifty-nine participants were not included in the analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine, Cytarabine + Idarubicin
Number analyzed (Participants) | 57
Months | 13.5 [1 to 23]

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Clofarabine, Cytarabine + Idarubicin
Serious Adverse Events (participants affected / at risk) | 36/59
Other Adverse Events (participants affected / at risk) | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Cytarabine + Idarubicin (N=59)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 19 (30)
Infection (Infections and infestations) | 17 (24)
Pain (General disorders) | 2 (3)
Renal Failure (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Headache (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Cytarabine + Idarubicin (N=59)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 19 (20)
Rash/hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 14 (14)
Mucositis/stomatitis (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 24 (25)
Vomiting (Gastrointestinal disorders) | 3 (3)
Febrile Neutropenia/fever of unknown origin (Infections and infestations) | 14 (16)
Infection (Infections and infestations) | 7 (7)
Elevated ALT/AST (Metabolism and nutrition disorders) | 11 (11)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Pain (Gastrointestinal disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes